CLINICAL TRIAL: NCT04750720
Title: Study of the Kinetics of COVID-19 Antibodies for 24 Months in Patients With Confirmed SARS-CoV-2 Infection According to the Clinical Severity of the Infection.
Brief Title: Study of the Kinetics of COVID-19 Antibodies for 24 Months in Patients With Confirmed SARS-CoV-2 Infection
Acronym: ABCOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Collaborators: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHRO-2020-12
Record Dates: First submitted 2021-02-09; First posted 2021-02-11 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Covid19; SARS-CoV-2
Keywords: Covid19; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Collection of biological samples (M0, M3, M6, M9, M12, M15, M18, M24) with associated data for the study of the kinetics of antibodies anti COVID-19 in subjects with documented SARS-CoV-2 infection (PCR and/or positive specific serology)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group with biological samples (Experimental): Collection of biological samples (M0, M3, M6, M9, M12, M15, M18, M24) with associated data for the study of the kinetics of antibodies anti COVID-19 in subjects with documented SARS-CoV-2 infection (PCR and/or positive specific serology). In the vaccine sub-study: additional blood and nasopharyngeal samples before and after vaccination, up to 6 months.
  Interventions: Other: Sampling by venipuncture (and eventually by nasopharyngeal swab)

INTERVENTIONS:
Other: Sampling by venipuncture (and eventually by nasopharyngeal swab) — Biological samples :
  * Serum and plasma from each donor for the purpose of performing (if applicable) the SARS-CoV-2 serologic test
  * PBMC (peripheral blood mononuclear cells)
  * Nasopharyngeal samples (not mandatory)
  Associated data :
  * Demographic data
  * Description of clinical manifestations related to SARS-CoV-2 infection
  * Notion of hospitalization/ambulatory follow-up
  Blood Fractioning
  * Serum and plasma aliquoted and stored under 250, 500 and 1000 µL (at -80°C)
  * Separation of PBMC on Lymphoprep and freezing in liquid nitrogen for subsequent analysis of immune system cells

SUMMARY:
The main objective of the study is to describe the temporal curve of COVID-19 IgG and neutralizing antibodies over 24 months in an identified population of patients who presented with SARS-CoV-2 virus infection. The secondary objectives are to characterize the kinetics of the antibodies according to the severity of the clinical presentation and patient's characteristics and to determine if the anti-SARS-CoV-2 antibodies retain their neutralizing capacity over time. A sub-study aims to describe the kinetic of neutralizing antibodies (in blood and nasal mucosa) after vaccination.

DETAILED DESCRIPTION:
Given the seriousness of the global health consequences of the COVID-19 pandemic and the difficulty of covering the world population with effective vaccination, several questions arise:

* Are the antibodies made by a patient neutralizing and do they protect the individual from further contamination?
* What is the persistence of the antibodies over time according to the clinical presentation, knowing that the very symptomatic forms have developed a much higher level of antibodies than the forms followed only on an outpatient basis and no less severe?
* What is the impact of vaccination (against wild-type virus and emerging variants) ? The investigators propose a single-center, observational study including 300 patients to answer the two questions, by selecting from the file of all the patients having had a positive RT-PCR 3 distinct groups: severe (hospitalized), pauci-symptomatic to moderate (followed in ambulatory only). Note: people living with HIV can be included in each of the groups.

MAIN EVALUATION

> Presence of specific anti-SARS-CoV-2 antibodies in the different study groups at M24 at each of the sampling times (M0, M3, M6, M9, M12, M15, M18, M24)

SECONDARY EVALUATION CRITERIA

* Presence of specific anti-SARS-CoV-2 antibodies in the different groups of the study at M12 and in each of the subgroups at M12 and M24
* Neutralizing capacity of anti-SARS-CoV-2 antibodies to M6, M12 and M24 on the classical strain and the new variants, before and after a possible vaccination against COVID-19
* Measurement of CD8 (CD38 + DR +), CD4 and activated B lymphocytes in culture This will make it possible to answer the question of the persistence or not of an immune response over 24 months, an essential element in the event of seasonal circulation of the virus in the years to come, and of the persistence or not of the neutralizing capacities of these antibodies in the over time, especially when the title approaches the detection threshold.

These information will be decisive in the event of successive waves of the SARS-CoV-2 epidemic given a low level of collective immunity (<10% in France at the end of 2020) in order to know whether previously affected patients are durably protected.

In the context of a lack of vaccine, results from this study would make it possible to select candidates for vaccination from the truly non-immune population.

Vaccine sub-study :

Study of the kinetic of neutralizing antibodies after vaccination :

Volunteers participants, provided they give a special agreement for the vaccine sub-study, will undergo an additional grid of samples to accurately study the kinetic of neutralizing antibodies before and monthly after (up to 6 months) receiving anti-SARS-CoV-2 vaccine (whatever the product used). A special attention will be given to the capacity of their antibodies to neutralize emerging variants. Samples will include blood and possibly nasopharyngeal swabs (not mandatory).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Having had a confirmed infection with CoV-2-SARS by RT-PCR and/or serology (IgM and/or IgG specific as significant)
* Being vaccinated against anti-SARS-CoV-2 (vaccine sub-study)
* Benefiting from a Social Security system
* Having consented to participate in the study
* Accepting regular follow-up for 24 months

Exclusion Criteria:

* Protected person (under guardianship or trusteeship)
* Person under the protection of justice
* Person unable to express consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
Presence of specific anti-SARS-CoV-2 antibodies | Month 0
  Presence of specific anti-SARS-CoV-2 antibodies in the different study groups at each sampling time
Presence of specific anti-SARS-CoV-2 antibodies | Month 3
  Presence of specific anti-SARS-CoV-2 antibodies in the different study groups at each sampling time
Presence of specific anti-SARS-CoV-2 antibodies | Month 6
  Presence of specific anti-SARS-CoV-2 antibodies in the different study groups at each sampling time
Presence of specific anti-SARS-CoV-2 antibodies | Month 9
  Presence of specific anti-SARS-CoV-2 antibodies in the different study groups at each sampling time
Presence of specific anti-SARS-CoV-2 antibodies | Month 12
  Presence of specific anti-SARS-CoV-2 antibodies in the different study groups at each sampling time
Presence of specific anti-SARS-CoV-2 antibodies | Month 15
  Presence of specific anti-SARS-CoV-2 antibodies in the different study groups at each sampling time
Presence of specific anti-SARS-CoV-2 antibodies | Month 18
  Presence of specific anti-SARS-CoV-2 antibodies in the different study groups at each sampling time
Presence of specific anti-SARS-CoV-2 antibodies | Month 24
  Presence of specific anti-SARS-CoV-2 antibodies in the different study groups at each sampling time

SECONDARY OUTCOMES:
Presence of specific anti-SARS-CoV-2 antibodies | Month 12
  Presence of specific anti-SARS-CoV-2 antibodies in the different study groups
Presence of specific anti-SARS-CoV-2 antibodies in subgroups | Month 12
  Presence of specific anti-SARS-CoV-2 antibodies in each of the subgroups
Presence of specific anti-SARS-CoV-2 antibodies in subgroups | Month 24
  Presence of specific anti-SARS-CoV-2 antibodies in each of the subgroups
Neutralizing capacity of anti-SARS-CoV-2 antibodies | Month 6
  Neutralizing capacity of anti-SARS-CoV-2 antibodies on the classical strain and the new variants, before and after a possible vaccination against COVID-19
Neutralizing capacity of anti-SARS-CoV-2 antibodies | Month 12
  Neutralizing capacity of anti-SARS-CoV-2 antibodies on the classical strain and the new variants, before and after a possible vaccination against COVID-19.
Neutralizing capacity of anti-SARS-CoV-2 antibodies | Month 24
  Neutralizing capacity of anti-SARS-CoV-2 antibodies on the classical strain and the new variants, before and after a possible vaccination against COVID-19.
Measurement of activated CD8 (CD38+DR+) in culture | Month 6
  Measurement of activated CD8 (CD38+DR+) in culture
Measurement of activated CD8 (CD38+DR+) in culture | Month 12
  Measurement of activated CD8 (CD38+DR+) in culture
Measurement of activated CD8 (CD38+DR+) in culture | Month 24
  Measurement of activated CD8 (CD38+DR+) in culture
Measurement of activated CD4 in culture | Month 6
  Measurement of activated CD4 in culture
Measurement of activated CD4 in culture | Month 12
  Measurement of activated CD4 in culture
Measurement of activated CD4 in culture | Month 24
  Measurement of activated CD4 in culture
Measurement of activated B lymphocytes in culture | Month 6
  Measurement of activated B lymphocytes in culture
Measurement of activated B lymphocytes in culture | Month 12
  Measurement of activated B lymphocytes in culture
Measurement of activated B lymphocytes in culture | Month 24
  Measurement of activated B lymphocytes in culture

CONTACTS AND LOCATIONS:
Overall Officials: Thierry PRAZUCK, MD, Principal Investigator — CHU Orléans
Locations (1):
- CHU Orléans, Orléans, France

REFERENCES:
- [Background] Corman VM, Landt O, Kaiser M, Molenkamp R, Meijer A, Chu DK, Bleicker T, Brunink S, Schneider J, Schmidt ML, Mulders DG, Haagmans BL, van der Veer B, van den Brink S, Wijsman L, Goderski G, Romette JL, Ellis J, Zambon M, Peiris M, Goossens H, Reusken C, Koopmans MP, Drosten C. Detection of 2019 novel coronavirus (2019-nCoV) by real-time RT-PCR. Euro Surveill. 2020 Jan;25(3):2000045. doi: 10.2807/1560-7917.ES.2020.25.3.2000045. PMID 31992387
- [Background] Rothan HA, Byrareddy SN. The epidemiology and pathogenesis of coronavirus disease (COVID-19) outbreak. J Autoimmun. 2020 May;109:102433. doi: 10.1016/j.jaut.2020.102433. Epub 2020 Feb 26. PMID 32113704
- [Background] Fafi-Kremer S, Bruel T, Madec Y, Grant R, Tondeur L, Grzelak L, Staropoli I, Anna F, Souque P, Fernandes-Pellerin S, Jolly N, Renaudat C, Ungeheuer MN, Schmidt-Mutter C, Collongues N, Bolle A, Velay A, Lefebvre N, Mielcarek M, Meyer N, Rey D, Charneau P, Hoen B, De Seze J, Schwartz O, Fontanet A. Serologic responses to SARS-CoV-2 infection among hospital staff with mild disease in eastern France. EBioMedicine. 2020 Sep;59:102915. doi: 10.1016/j.ebiom.2020.102915. Epub 2020 Jul 31. PMID 32747185
- [Derived] Bolland W, Michel V, Planas D, Hubert M, Staropoli I, Guivel-Benhassine F, Porrot F, N'Debi M, Rodriguez C, Fourati S, Prot M, Planchais C, Hocqueloux L, Simon-Loriere E, Mouquet H, Prazuck T, Pawlotsky J-M, Bruel T, Schwartz O, Buchrieser J. High fusion and cytopathy of SARS-CoV-2 variant B.1.640.1. J Virol. 2024 Jan 23;98(1):e0135123. doi: 10.1128/jvi.01351-23. Epub 2023 Dec 13. PMID 38088562
- [Derived] Clairon Q, Prague M, Planas D, Bruel T, Hocqueloux L, Prazuck T, Schwartz O, Thiebaut R, Guedj J. Modeling the kinetics of the neutralizing antibody response against SARS-CoV-2 variants after several administrations of Bnt162b2. PLoS Comput Biol. 2023 Aug 7;19(8):e1011282. doi: 10.1371/journal.pcbi.1011282. eCollection 2023 Aug. PMID 37549192
- [Derived] Garcia L, Woudenberg T, Rosado J, Dyer AH, Donnadieu F, Planas D, Bruel T, Schwartz O, Prazuck T, Velay A, Fafi-Kremer S, Batten I, Reddy C, Connolly E, McElheron M, Kennelly SP, Bourke NM, White MT, Pelleau S. Kinetics of the SARS-CoV-2 Antibody Avidity Response Following Infection and Vaccination. Viruses. 2022 Jul 8;14(7):1491. doi: 10.3390/v14071491. PMID 35891471